CLINICAL TRIAL: NCT00306332
Title: T-cel and B-cell Depletion in Allogeneic Peripheral Blood Stem Cell Transplantation by Using Immunomagnetic Negative and Positive Selection Procedures
Brief Title: T-cell and B-cell Depletion in Allogeneic Peripheral Blood Stem Cell Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis has shown that the objectives of this study can not be reached
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSCT10
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Leukemia, Myeloid; Leukemia, Lymphocytic; Myelodysplastic Syndrome; Leukemia, Myeloid, Chronic; Lymphoma
Keywords: Allogeneic Stem cell transplantation; T-cell depletion; B-cell depletion; Immunomagnetic selection
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Lymphoid; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma

INTERVENTIONS:
Procedure: T-cell and B-cell depletion

SUMMARY:
T-cell and B-cell depletion in allogeneic peripheral blood stem cell transplantation by using immunomagnetic negative and positive selection procedures

Background:

Removal of T-cells from the donor graft (T-cell depletion) offers the possibility for prevention of GVHD and subsequently less transplant related morbidity and mortality after allogeneic stem cell transplantation (SCT). There are several techniques to deplete T-cells from the stem cell grafts e.g. physical, immunological and combined physical / immunological separation methods. All these techniques result in a stem cell graft with sufficient CD34+ stem cells combined with an adequate depletion of T and B cells. CD34+ selected stem cell grafts are very pure and do not contain any additional cell populations. In contrast, CD3+/CD19+ depleted grafts still contain NK-cells, monocytes and dendritic cells that are part of the innate immune system. Theoretically,the presence of these cells may positively influence immunological reconstitution and the graft-versus-leukaemia (GVL) effect, respectively, resulting in improved outcome after SCT

Objectives:

To evaluate the differences in immunological reconstitution, transplant related mortality, disease-free survival and overall survival after T-cell depleted allogeneic SCT for haematological malignancies using either immunomagnetic CD34+ selection or immunomagnetic CD3+/CD19+ depletion using the CliniMACS system in approximately 270 consecutive patients.

Additionally in this study in 20 consecutive patients the kinetics of NK-cel reconstitution and differences in NK-cell repertoire will be monitored. NK-cell mediated anti-tumor reactivity will be monitored in patients transplanted with and without NK-cells in the stem cell graft (CD3+/CD19+ depletion, versus CD34+ selection). Secondary objectives are to evaluate the clinical relevance of minor histocompatibility-specific cytotoxic T-cell responses for the GVL effect, the kinetics of NK-cell reconstitution and differences in NK-cell repertoire using the different T-cell depletion protocols.

Design:

Single center prospective randomised phase III study

Population:

Patients eligible for allogeneic SCT according to the standard criteria of our institution who will receive an allogeneic T- and B-cell depleted SCT with peripheral stem cells of an HLA-identical sibling donor or an HLA-identical unrelated voluntary (VUD) donor.

Intervention:

T-cell depletion will be conducted using two different techniques: either immunomagnetic CD34+ selection or immunomagnetic CD3+/CD19+ depletion.

Endpoints:

Primary endpoints are immunological reconstitution, relapse, disease free survival and overall survival. Secondary endpoints: NK-cell reconstitution and NK-cell mediated anti-tumour reactivity. Cytotoxic T-cell responses for the GVL effect.

Estimated efforts and risks for participating patients:

We don't expect any extra patient efforts or risks because T-cell depletion is a standard procedure in our clinic for many years. There is extensive experience with immunological T-cell depletion techniques. We hypothesize CD3+/CD19+ depletion will favour stem cell transplant outcome. Immunological and molecular biological studies will be performed on blood samples already obtained as part of the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of:

  * De novo acute myeloid leukaemia in first or second remission.
  * Secondary acute myeloid leukaemia in first or second remission supervening after myelodysplastic syndrome or cytotoxic / immunosuppressive therapy.
  * Acute lymphoblastic leukaemia in first or second remission.
  * Myelodysplastic syndrome.
  * Chronic myeloid leukaemia, patients who are candidate for SCT.
  * Malignant lymphoma following relapse or first line therapy resistant.
  * Aggressive mantle cell lymphoma in first complete remission.
* Age 18-65 years.
* WHO performance 0-1 (see appendix ).
* Availability of an HLA-identical sibling or HLA, A, B, DRB, DQB -identical VUD donor.
* Life expectancy > 3 months.
* Witnessed written informed consent.

Exclusion Criteria:

* Patients with severe cardiac dysfunction (NYHA-classification II-IV)
* Patients with severe pulmonary dysfunction (vital capacity or diffusion < 70% of predicted value).
* Patients with hepatic dysfunction, bilirubin or transaminases > 2.5 x upper normal limit
* Patients with renal dysfunction, serum creatinin > 150 umol/liter or clearance < 40 ml/minute.
* Patients with a history of moderate ore severe CNS disturbances and psychiatric problems.
* Prior treatment with chemotherapy, immunotherapy, radiation therapy or surgery within the last 3 weeks before entering the study.
* Patients with active uncontrolled infections.
* Patients who are poor medical risks because of non malignant systemic disease.
* Patients with severe coagulopathy.
* Patients to be known HIV positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
relapse
event-free survival
survival

SECONDARY OUTCOMES:
clinical relevance of mHag-specific CTL responses for the GVL effect
Kinetics of NK-cel reconstitution
Differences in NK-cell repertoire
NK cell mediated anti tumor reactivity

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Schaap, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- 476 Hematology, University Medical Centre St Radboud Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Background] Schaap N, Schattenberg A, Bar B, Preijers F, Geurts van Kessel A, van der Maazen R, de Boo T, de Witte T. Outcome of transplantation for standard-risk leukaemia with grafts depleted of lymphocytes after conditioning with an intensified regimen. Br J Haematol. 1997 Sep;98(3):750-9. doi: 10.1046/j.1365-2141.1997.d01-3499.x. PMID 9332335
- [Background] Schattenberg A, Schaap N, Preijers F, van der Maazen R, de Witte T. Outcome of T cell-depleted transplantation after conditioning with an intensified regimen in patients aged 50 years or more is comparable with that in younger patients. Bone Marrow Transplant. 2000 Jul;26(1):17-22. doi: 10.1038/sj.bmt.1702451. PMID 10918401
- [Background] Schaap N, Schattenberg A, Bar B, Preijers F, van de Wiel van Kemenade E, de Witte T. Induction of graft-versus-leukemia to prevent relapse after partially lymphocyte-depleted allogeneic bone marrow transplantation by pre-emptive donor leukocyte infusions. Leukemia. 2001 Sep;15(9):1339-46. doi: 10.1038/sj.leu.2402203. PMID 11516094